CLINICAL TRIAL: NCT01271855
Title: CRAMPS Trial: Controlled Randomized Trial Assessing Maternal Post-partum Pain With Suppositories
Brief Title: Assessing Maternal Post-partum Pain With Suppositories
Acronym: CRAMPS
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Loyola University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 201720
Record Dates: First submitted 2011-01-05; First posted 2011-01-07 (Estimated); Results first posted 2018-02-06 (Actual); Last update posted 2018-03-07 (Actual); Status verified 2018-02

CONDITIONS: Pain
Keywords: Belladonna; Opium; Suppository
MeSH Terms: conditions — Pain

STUDY DESIGN:
Intervention Model Description: Participants will be randomized to receive either a belladonna and opioid suppository or a glycerin suppository (placebo) every eight hours after delivery during the first 24 hours after delivery using a 1:1 allocation
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Glycerin suppository (Placebo Comparator): Women assigned to this arm receive a glycerin suppository (placebo) every 8 hours after delivery during the first 24 hours postpartum
  Interventions: Drug: Glycerin Suppository
- Belladonna and opioid suppository (Experimental): Women assigned to this arm receive a belladonna and opioid (B&O) suppository every 8 hours after delivery during the first 24 hours postpartum
  Interventions: Drug: Belladonna and opioid suppository

INTERVENTIONS:
Drug: Belladonna and opioid suppository — Belladonna and opioid suppository 16.2mg/30mg per rectum every 8 hours for 24 hours following delivery
  Arms: Belladonna and opioid suppository
Drug: Glycerin Suppository — A vegetable oil suppository (placebo) per rectum every 8 hours for the first 24 hours following delivery.
  Arms: Glycerin suppository

SUMMARY:
This trial will evaluate whether the routine use of belladonna/opium (B&O) suppositories improve patients' self-reported pain control in the first 24-hours after delivery.

DETAILED DESCRIPTION:
Childbirth is commonly regarded as one of life's most painful experiences and, like childbirth, the postpartum period can also be painful for women. Pain in the immediate postpartum period may significantly affect a woman's overall delivery experience. Pain control is especially important in this period, as women are bonding with their infant and trying to initiate breastfeeding, which may be adversely affected by poor pain management.

Postpartum pain may come from multiple sources. Women experience uterine cramping as a result of uterine involution. Depending on delivery type, women may also have incision pain following cesarean section or perineal pain resulting from episiotomy, perineal tears, or generalized genital trauma during delivery. Perineal pain is common, present in 75% of patients with intact perineum and up to 95-97% with perineal lacerations or episiotomies during the first day after delivery. Commonly employed methods of controlling postpartum pain include opioid analgesics, non-steroidal anti-inflammatories, acetaminophen, and topical analgesics. Pain medication is generally administered via oral or intravenous route. Several studies have investigated suppositories as an alternative method of improving pain following delivery. A double-blinded randomized controlled trial by Wilasrusmee et al (2008) showed naproxen suppositories to be effective for reducing perineal pain after vaginal delivery. Another study showed prophylactic rectal diclofenac to provide effective analgesia after perineal repair, maintained into second and third day postpartum, and a Cochrane Review showed NSAID suppositories to be associated with less pain 24 hours after birth.

Rectal analgesia provides a means of improving pain control through local effects on the perineum and uterus while possibly decreasing systemic absorption, which may in turn decrease systemic side effects and transmission to the newborn infant through breast milk. B&O suppositories contain two medications that could potentially decrease postpartum pain. Morphine, the principle agent in opium, binds opioid receptors and blocks ascending pain pathways. Atropine, a major active component of belladonna, blocks acetylcholine receptors, leading to smooth muscle relaxation. This quality may significantly improve pain from uterine contractions during the postpartum period. The primary aim of our study is to investigate whether belladonna and opium suppositories decrease patient-reported pain in the immediate postpartum period.

ELIGIBILITY:
Inclusion Criteria:

* Anticipated Vaginal or Cesarean delivery at Gottlieb Medical Center or Loyola University Medical Center
* > 34 weeks gestation at time of delivery
* > 18 years old
* No known allergy to belladonna, opium, or vegetable oil suppositories
* Able to consent and complete study documents

Exclusion Criteria:

* Chronic pain condition or on narcotic medication prior to admission
* Contraindications to B&O suppositories, including patients with glaucoma, severe hepatic, or renal disease; bronchial asthma; narcotic idiosyncrasies; respiratory depression; convulsive disorders; acute alcoholism; delirium tremens; history of hypersensitivity to any component of product.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2009-07-22 (Actual); Primary Completion 2011-09-29 (Actual); Study Completion 2011-09-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kimberly Kenton, M.D., Principal Investigator — Northwestern University
Locations (2):
- United States (2):
  - Loyola Univeristy Medical Center, Maywood, Illinois
  - Gottlieb Memorial Hospital, Melrose Park, Illinois

IPD SHARING:
Plan to Share IPD: No
There is no plan to share individual participant data.

REFERENCES:
- [Background] Macarthur AJ, Macarthur C. Incidence, severity, and determinants of perineal pain after vaginal delivery: a prospective cohort study. Am J Obstet Gynecol. 2004 Oct;191(4):1199-204. doi: 10.1016/j.ajog.2004.02.064. PMID 15507941
- [Background] Wilasrusmee S, Chittachareon A, Jirasiritum S, Srisangchai P. Naproxen suppository for perineal pain after vaginal delivery. Int J Gynaecol Obstet. 2008 Jul;102(1):19-22. doi: 10.1016/j.ijgo.2008.01.015. Epub 2008 Mar 5. PMID 18321517
- [Background] Searles JA, Pring DW. Effective analgesia following perineal injury during childbirth: a placebo controlled trial of prophylactic rectal diclofenac. Br J Obstet Gynaecol. 1998 Jun;105(6):627-31. doi: 10.1111/j.1471-0528.1998.tb10177.x. PMID 9647153
- [Background] Hedayati H, Parsons J, Crowther CA. Rectal analgesia for pain from perineal trauma following childbirth. Cochrane Database Syst Rev. 2003;(3):CD003931. doi: 10.1002/14651858.CD003931. PMID 12917995
- [Background] Gallagher EJ, Bijur PE, Latimer C, Silver W. Reliability and validity of a visual analog scale for acute abdominal pain in the ED. Am J Emerg Med. 2002 Jul;20(4):287-90. doi: 10.1053/ajem.2002.33778. PMID 12098173
- [Background] Bijur PE, Silver W, Gallagher EJ. Reliability of the visual analog scale for measurement of acute pain. Acad Emerg Med. 2001 Dec;8(12):1153-7. doi: 10.1111/j.1553-2712.2001.tb01132.x. PMID 11733293
- [Background] DeLoach LJ, Higgins MS, Caplan AB, Stiff JL. The visual analog scale in the immediate postoperative period: intrasubject variability and correlation with a numeric scale. Anesth Analg. 1998 Jan;86(1):102-6. doi: 10.1097/00000539-199801000-00020. PMID 9428860
- [Derived] Deussen AR, Ashwood P, Martis R, Stewart F, Grzeskowiak LE. Relief of pain due to uterine cramping/involution after birth. Cochrane Database Syst Rev. 2020 Oct 20;10(10):CD004908. doi: 10.1002/14651858.CD004908.pub3. PMID 33078388

RESULTS

PARTICIPANT FLOW:
Recruitment Details: For this study, participants were recruited between August 1, 2009 and October 1, 2011 (26 months)
Groups:
- Glycerin Suppository: Women assigned to this arm receive a vegetable oil suppository (placebo) per rectum every 8 hours for the first 24 hours following delivery.
- Belladonna and Opioid Suppository: Women assigned to this arm receive a Belladonna and opioid suppository 16.2mg/30mg per rectum every 8 hours for 24 hours following delivery
Period: Overall Study
Arm/Group | Glycerin Suppository | Belladonna and Opioid Suppository
Started | 48 | 52
Completed | 48 | 52
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Glycerin Suppository | Belladonna and Opioid Suppository | Total
Number analyzed (Participants) | 48 | 52 | 100
Age, Continuous [Mean (Standard Deviation); unit: years] | 29.40 (5.78) | 29.29 (5.76) | 29.34 (5.74)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 48 | 52 | 100
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 17 | 19 | 36
  Not Hispanic or Latino | 24 | 22 | 46
  Unknown or Not Reported | 7 | 11 | 18
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 0 | 1 | 1
  Black or African American | 7 | 6 | 13
  White | 24 | 25 | 49
  Other Race | 2 | 7 | 9
  Unknown or Not Reported | 15 | 13 | 28
Region of Enrollment [Number; unit: participants]
  United States | 48 | 52 | 100
Gravidity [Median (Inter-Quartile Range); unit: Count of pregnancies] | 2.5 [2 to 3] | 2 [1 to 3] | 2 [2 to 3]
Parity [Median (Inter-Quartile Range); unit: Pregnancies to a viable gestational age] — Population: The parity count for one participant in the Belladonna and opioid suppository group is unknown
  Pregnancies to a viable gestational age
    number analyzed (Participants) | 48 | 51 | 99
    (all) | 1 [1 to 2] | 1 [0 to 2] | 1 [0 to 2]
Gestational Age [Mean (Standard Deviation); unit: Weeks] — Population: The gestational age for one participant in the Belladonna and opioid suppository group is unknown, and the gestational age for one participant in the Glycerin suppository group is unknown
  Weeks
    number analyzed (Participants) | 47 | 51 | 98
    (all) | 38.68 (1.24) | 39.09 (1.05) | 38.89 (1.16)
Route of Delivery [Count of Participants; unit: Participants]
  Normal spontaneous vaginal delivery (NSVD) | 31 | 42 | 73
  Cesarean | 17 | 10 | 27
Breastfeeding [Count of Participants; unit: Participants]
  Breastfeeding | 37 | 41 | 78
  Not Breastfeeding | 8 | 9 | 17
  Breastfeeding is unknown or not reported | 3 | 2 | 5
Visual Analogue Scale Pain Score [Median (Inter-Quartile Range); unit: units on a scale] — Patients' baseline Visual Analog Scale (VAS) pain score was recorded at 0 hours after delivery. This scale ranges from 0 to 10 (0=no pain and 10=worst pain). Population: The baseline visual analogue pain score for two participants in the Belladonna and opioid suppository group is unknown, and the baseline visual analogue pain score for one participant in the Glycerin suppository group is unknown
  units on a scale
    number analyzed (Participants) | 47 | 50 | 97
    (all) | 0 [0 to 2] | 0 [0 to 4] | 0 [0 to 4]

OUTCOME MEASURES:

1. Primary Outcome: Pain Level Twenty Four Hours After Delivery
Description: The primary outcome is pain measured at 24-hours after delivery. Patients will be asked to report a Visual Analog Scale (VAS) pain score at 24-hours after delivery. This scale ranges from 0 to 10 (0=no pain and 10=worst pain).
Time Frame: Twenty-four hours
Population: The 24-hour visual analogue pain score for two participants in the Belladonna and opioid suppository group is unknown, and the 24-hour visual analogue pain score for one participant in the Glycerin suppository group is unknown
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Glycerin Suppository | Belladonna and Opioid Suppository
Number analyzed (Participants) | 47 | 50
units on a scale | 1 [0 to 3] | 2 [0 to 3]
Statistical Analysis 1: Comparison: Glycerin Suppository vs Belladonna and Opioid Suppository; The null hypothesis is that there is no difference in the visual analogue pain score scale (VAS) between participants in the Glycerin suppository group and those in the Belladonna and opioid suppository group 24-hours after delivery; Test type: Superiority; p = .35, Wilcoxon (Mann-Whitney); Z-Score = 0.93 — The z-score is a standardized version of the Wilcoxon test statistic. In this study, z-scores with an absolute value exceeding 1.96 signal the two groups have meaningfully different pain scores. Other values would fail to reject the null hypothesis

2. Secondary Outcome: Number of Patients Taking Additional Pain Medications
Description: Twenty-four hours after delivery, the number of participants taking additional pain medications will be recorded.
Time Frame: Twenty-four hours
Measure: Count of Participants; unit: Participants
Arm/Group | Glycerin Suppository | Belladonna and Opioid Suppository
Number analyzed (Participants) | 48 | 52
Participants
  Taking additional pain medications | 40 | 47
  Not taking additional pain medications | 8 | 5
Statistical Analysis 1: Comparison: Glycerin Suppository vs Belladonna and Opioid Suppository; The null hypothesis is that there is no difference in the odds of taking additional pain medications between participants in the Glycerin suppository group and those in the Belladonna and opioid suppository group 24-hours after delivery; Test type: Superiority; p = .30, Regression, Logistic; Odds Ratio (OR) = 1.88, 95% CI 2-sided [0.57 to 6.21]

3. Secondary Outcome: Patient Satisfaction
Description: Patients' satisfaction with their pain control is recorded at the time of discharge using a five point scale ranging from 1 (Not Satisfied) to 3 (Okay) to 5 (Very Satisfied).
Time Frame: Discharge
Population: The pain satisfaction at discharge score is unknown for eight participants in the Belladonna and opioid suppository group, and the pain satisfaction at discharge score is unknown for six participants in the Glycerin suppository group.
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Glycerin Suppository | Belladonna and Opioid Suppository
Number analyzed (Participants) | 42 | 44
units on a scale | 4 [3 to 5] | 5 [3 to 5]
Statistical Analysis 1: Comparison: Glycerin Suppository vs Belladonna and Opioid Suppository; The null hypothesis is that there is no difference in the pain satisfaction score between participants in the Glycerin suppository group and those in the Belladonna and opioid suppository group at discharge; Test type: Superiority; p = .02, Wilcoxon (Mann-Whitney); Z-Score = 2.34 — The z-score is a standardized version of the Wilcoxon test statistic. In this study, z-scores with an absolute value exceeding 1.96 signal the two groups have meaningfully different satisfaction scores. Other values fail to reject the null hypothesis

ADVERSE EVENTS:
Time Frame: Adverse event data were collected for 28 months
Arm/Group | Glycerin Suppository | Belladonna and Opioid Suppository
All-Cause Mortality (participants affected / at risk) | 0/48 | 0/52
Serious Adverse Events (participants affected / at risk) | 0/48 | 0/52
Other Adverse Events (participants affected / at risk) | 22/48 | 23/52
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Glycerin Suppository (N=48) | Belladonna and Opioid Suppository (N=52)
Dry Mouth (Gastrointestinal disorders) | 12 (12) | 19 (19)
Difficulty Urinating (Renal and urinary disorders) | 2 (2) | 3 (3)
Sensitivity to Light (Eye disorders) | 0 (0) | 1 (1)
Tachycardia (Cardiac disorders) | 0 (0) | 2 (2)
Dizziness (General disorders) | 6 (6) | 3 (3)
Blurred Vision (Eye disorders) | 1 (1) | 1 (1)
Constipation (Gastrointestinal disorders) | 3 (3) | 3 (3)
Nausea (General disorders) | 5 (5) | 8 (8)
Emesis (General disorders) | 2 (2) | 2 (2)
Itching (Skin and subcutaneous tissue disorders) | 6 (6) | 4 (4)
Headache (General disorders) | 1 (1) | 2 (2)
Tinnitus (Ear and labyrinth disorders) | 1 (1) | 0 (0)

LIMITATIONS AND CAVEATS:
There are no limitations or caveats to report

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No